CLINICAL TRIAL: NCT06114589
Title: An Observational Study to Develop Molecular Integrated Predictive Models of Breast Radio-toxicity (Precise-RTox)
Brief Title: A Study to Develop Molecular Integrated Predictive Models of Breast Radio-toxicity (Precise-RTox)
Acronym: (Precise-RTox)
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2022-29
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast radiation treatment is burdened by acute and chronic toxicities, in most cases mild. However, considering the excellent life expectancy of patients with breast cancer, maintaining a low toxicity profile is of primary importance in order to guarantee a satisfactory quality of life. The definition of the molecular and genetic variables related to radiotoxicity and their integration into predictive molecular signatures may allow the risk of toxicity to be individualized. This would provide the clinician with a useful tool in order to personalize the radiation treatment, thus being able to choose the best technique or schedule for each patient.

DETAILED DESCRIPTION:
Breast radiation treatment is burdened by acute and chronic toxicities, in most cases mild. However, considering the excellent life expectancy of patients with breast cancer, maintaining a low toxicity profile is of primary importance in order to guarantee a satisfactory quality of life. Currently there are numerous predictive models of toxicity (Normal Tissue Complication Probability, NTCP) which are based on dosimetric and sometimes also clinical data. To date, they do not include individual genetic variability. However, it is believed that inter-individual variability may be responsible for up to 40% of actinic toxicity. Multiparametric models that consider genetics, dose and clinical aspects probably better reflect the complexity of radiotoxicity than models that rely on a single parameter and it is possible to integrate such parameters using a machine learning approach. The definition of the molecular and genetic variables related to radiotoxicity and their integration into predictive molecular signatures would therefore allow the risk to be individualized. This would provide the clinician with a useful tool in order to personalize the radiation treatment, thus being able to choose the best technique or schedule for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Ability to express appropriate informed consent to treatment;
* Distant nonmetastatic breast cancer;
* Histology: infiltrating NST(no special type)/lobular carcinoma or ductal carcinoma in situ;
* Stage: pTis; pT1-3 pN1-3 M0;
* Hormone receptors, HER-2 status: Any;
* Breast-conserving surgery. Both the sentinel lymph node biopsy and axillary lymphadenectomy. Negative surgical margins.
* Candidates for postoperative radiation treatment.

Exclusion Criteria:

* Refusal of radiotherapy treatment (i.e., absence of signed informed consent);
* Previous radiation therapy at the same site;
* Concomitant chemotherapy with anthracyclines or taxanes;
* Inability to maintain treatment position;
* Partial breast radiotherapy (PBI);
* Male breast cancer;
* Mastectomy surgery.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with distant non-metastatic breast cancer candidated to radiotherapy after conservative surgery
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Generation of a predictive model for actinic fibrosis. | up to 2 years after start of treatment
  Identification of a predictive model of actinic fibrosis in the breast, with sensitivity of at least 75% and specificity of 90%. Fibrosis is defined as grade ≥2 (CTCAE v 4.0) or skin induration as grade ≥2 defined according to CTCAE v 4.0 .

SECONDARY OUTCOMES:
Generation of a predictive model for acute skin toxicity | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict acute skin toxicity defined according to CTCAE scale v4.0 as dermatitis grade ≥2 or ulceration of the skin of grade ≥2
Generation of a predictive model for late skin toxicity | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict late skin toxicity defined according to CTCAE scale v4.0 as grade 2 telangiectasia or grade 2 hyperpigmentation
Generation of a predictive model for acute pain | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict acute pain of grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for chronic pain | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict chronic pain grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for fatigue | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict fatigue of grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for lymphedema | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict ipsilateral limb lymphedema of grade ≥2 defined according to CTCAE v4.0
Generation of a predictive model for hypothyroidism | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict hypothyroidism of grade ≥2 defined according to CTCAE v4.0
Generation of a predictive model for contra-lateral breast cancer | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict secondary neoplasia to the contra-lateral breast according to CTCAE v4.0
Generation of a predictive model for cardiotoxicity | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict cardiotoxicity defined as reduction at echocardiography of Global Longitudinal Strain (GLS) ≥10% compared to baseline
Generation of a predictive model for cardiotoxicity | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict grade ≥2 cardiovascular events defined according to CTCAE v4.0
Generation of a predictive model for aesthetic outcome | up to 2 years after start of treatment
  Sensitivity of a model combining different variables to predict aesthetic outcome defined as fair/poor, according to Harvard score
Generation of a predictive model for acute skin toxicity | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict acute skin toxicity defined according to CTCAE scale v4.0 as dermatitis grade ≥2 or ulceration of the skin of grade ≥2
Generation of a predictive model for late skin toxicity | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict late skin toxicity defined according to CTCAE scale v4.0 as grade 2 telangiectasia or grade 2 hyperpigmentation
Generation of a predictive model for acute pain | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict acute pain of grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for chronic pain | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict chronic pain of grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for fatigue | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict fatigue of grade ≥2 defined according to CTCAE scale v4.0
Generation of a predictive model for lymphedema | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict ipsilateral limb lymphedema of grade ≥2 defined according to CTCAE v4.0
Generation of a predictive model for hypothyroidism | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict hypothyroidism of grade ≥2 defined according to CTCAE v4.0
Generation of a predictive model for contra-lateral breast cancer | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict secondary neoplasia to the contra-lateral breast according to CTCAE v4.0
Generation of a predictive model for cardiotoxicity | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict cardiotoxicity defined as reduction at echocardiography of Global Longitudinal Strain (GLS) ≥10% compared to baseline
Generation of a predictive model for cardiotoxicity | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict grade ≥2 cardiovascular events defined according to CTCAE v4.0
Generation of a predictive model for aesthetic outcome | up to 2 years after start of treatment
  Specificity of a model combining different variables to predict aesthetic outcome defined as fair/poor, according to Harvard score
Comparison between toxicity risk in treatment plans using protons or photons | up to 2 years after start of treatment
  Difference in frequency of high risk toxicity between treatment plans using protons or photons

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Vinante, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Barbara Belletti, PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy